# PROJECT TITLE

Mindfulness-Based Cognitive Therapy Delivered via Group Videoconferencing for Acute Coronary Syndrome Patients with Elevated Depression Symptoms

### **Version Date**

March 31, 2021

## NCT Number

03878160

#### **DATA ANALYSIS**

#### Focus groups

Focus groups will be audio recorded, transcribed, and iteratively analyzed using thematic content analysis in NVivo 11. With mentorship from study staff, the RA and PI will separately review each transcript to identify common themes and develop a coding framework. We will review our results for agreement and comparison to the raw data, and resolve discrepancies through discussion with study staff until reliability is reached (Kappa>.80).

#### **Survey Measures**

The following measures will be used to assess depression symptoms, trait mindfulness, health behaviors, and other psychological, behavioral, and physical constructs that may potentially be impacted by the MBCT intervention in subsequent trials: Five Factor Mindfulness Questionnaire15 item (FFMQ-15), Perceived Stress Scale-4 (PSS-4), Difficulties in Emotion Regulation Scale (DERS), Positive Affect Negative Affect Schedule (PANAS), Rumination Response Scale (RRS), Inclusion of Other in Self Scale (SOFI), Interpersonal Reactivity Index (IRI), Dispositional Positive Emotions Scale- Compassion (DPES-C), Medical Outcomes Study – Specific Adherence Scale (MOS- SAS), PROMIS- Physical Function, PHQ-9, and SF-12. We will explore descriptive statistics (e.g., medians and interquartile ranges).